CLINICAL TRIAL: NCT03206398
Title: Influence of an Anti-gravity Treadmill on Functional Outcome in Non-operatively Treated Pelvic Fractures - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. med. Ralf Henkelmann, PI, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1007
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Weight-bearing; Rehabilitation

STUDY DESIGN:
Intervention Model Description: anti-gravity treadmill for a total of 40 days in addition to physiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pelvic fracture (Other): patients with pelvic fracture will additionally be treated with anti-gravity treadmill
  Interventions: Device: anti-gravity treadmill

INTERVENTIONS:
Device: anti-gravity treadmill — anti-gravity treadmill for a total of 40 days in addition to physiotherapy

SUMMARY:
Non-operative treatment of pelvic fractures is possible. Immobilisation implies different adjustment processes. Patients with pelvic ring fractures and partial weight bearing have to obtain theses. The aim of this pilot study was to prove the additional effect of the anti-gravity treadmill in patients with non-operatively treated pelvic fractures.

DETAILED DESCRIPTION:
We prospectively included patients with non-operatively treated pelvic fractures as the intervention group (IG) and healthy volunteers of different age, sex and body mass index (BMI) as the reference group (RG).

Patients of the IG participated in a training session every three days with an anti-gravity treadmill (Picture 1, alterG®, www.alterg.com) for a total of 40 days in addition to physiotherapy, lymph drainage massage and manual therapy.

Patients were evaluated on three successive dates: Baseline (S1), after mobilization without crutches with full weight-bearing (20 days, S2) and after 40 days (S3)

ELIGIBILITY:
Inclusion Criteria:

* patients with non-operatively treated pelvic fractures

Exclusion Criteria:

* pregnancy, neuromuscular disorders, preexisting muscle atrophy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
standardized gait analysis | Day 1 - 40 days
  standardized gait analysis was done with fluorescent markers and two cameras

SECONDARY OUTCOMES:
numeric rating scale | Day 1 - 40 days
  numeric rating scale (NRS) to evaluate pain
dynamic gait index | Day 1 - 40 days
  rated gait index validated

IPD SHARING:
Plan to Share IPD: Undecided